CLINICAL TRIAL: NCT03158363
Title: A New Model of Acute Febrile Disease - Combining Endotoxemia, Immobilisation and Fasting in Healthy Young Males.
Brief Title: A New Model of Acute Febrile Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TheValidationStudy
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2017-05

CONDITIONS: Immobilization, Tonic; Fasting; Endotoxemia; Metabolism
Keywords: immobilization; fasting; endotoxemia; LPS; metabolism; model of disease
MeSH Terms: conditions — Immobility Response, Tonic; Fasting; Endotoxemia | interventions — Lipopolysaccharides; Immobilization

STUDY DESIGN:
Intervention Model Description: Healthy young adults will be randomized to either intervention "Endotoxemia, 36 hour immobilization and fasting" or "overnight fast" being the control day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "LPS, 36 hour immobilization and fast" (Experimental): Interventions:
  Test subjects undergo 48 hour exercise restriction and overnight fast.
  Study day 1:
  - LPS (1 ng/kg) will be administered. Test subjects will fast and bedrest for the rest of the study period.
  Study day 2:
  * 3 hour Basal period: Continued fast and bedrest. Phenylalanine, tyrosine, carbamide, glucose and palmitate tracers are infused. Muscle and fat biopsies are taken from m. vastus lateralis and stomach.
  * 3 hour hyperinsulinemic euglycemic clamp period with muscle and fat biopsies.
  Study day 3:
  - Blood sample.
  Interventions: Other: LPS, 36 hour immobilization and fast
- "Control" (No Intervention): Test subjects undergo overnight fast. No exercise restrictions.
  * 3 hour Basal period: Continued fast and bedrest. Phenylalanine, tyrosine, carbamide, glucose and palmitate tracers are infused. Muscle and fat biopsies are taken from m. vastus lateralis and stomach.
  * 3 hour hyperinsulinemic euglycemic clamp period with muscle and fat biopsies.

INTERVENTIONS:
Other: LPS, 36 hour immobilization and fast — LPS endotoxin is administered on study day 1 and immobilization and fast continue throughout study day 1 and 2.
  Arms: "LPS, 36 hour immobilization and fast"

SUMMARY:
The investigators want to establish a new model of acute febrile disease by mimicking the conditions seen in hospitalized patients in regards to inflammation, immobilisation and fasting. In this new model of disease, healthy young adults will be given lipopolysaccharide (LPS) to induce endotoxemia and inflammation/fever and then fast and bedrest for 36 hours. Glucose, fat and protein metabolism will be investigated using clamp technique and tracer methodology together with intracellular signalling pathway activation in muscle and fat biopsies. This new model of disease will later be used in another study to investigate different protein supplement´s effect on muscle waste during acute febrile disease.

DETAILED DESCRIPTION:
The investigators want to establish a new model of acute febrile disease by mimicking the conditions seen in hospitalized patients in regards to inflammation, immobilisation and fasting. In this new model of disease, healthy young adults will be given lipopolysaccharide (LPS) to induce endotoxemia and inflammation on study day 1 and then fast and bedrest for 36 hours (Study day 2). Glucose, fat and protein metabolism will be investigated using clamp technique and tracer methodology together with intracellular signalling pathway activation in muscle and fat biopsies. This new model of disease will later be used in another study to investigate different protein supplement´s effect on muscle waste during acute febrile disease.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* 20 < BMI < 30
* 20 < Age < 40 years
* Written consent prior to trial

Exclusion Criteria:

* Participation in trials using ionized radiation a year prior to this trial.
* Comprehensive x-ray examinations in the study period.
* In case of immobilization of an extremity, the extremity should be fully re- habilitated and this should be stated by a physician or physiotherapist. The test subject's word for this will be sufficient.
* Allergies to eggs or soy oil.
* Diseases: Diabetes, epilepsy, ongoing infectious disease, immunodeficiency, heart disease, dysregulated hypertension.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | After a 3 hour clamp
  Measured by hyperinsulinemic euglycemic clamp technique

SECONDARY OUTCOMES:
Protein metabolism | measured at baseline and after 3 hours of clamp
  Quantified by phenylalanine and tyrosine tracer methodology (whole body and the forearm model)
ketone body metabolic changes | measured at baseline and after 3 hours of clamp
  measurement of ketone bodies
inflammation | measurements over 36 hours
  Quantified by C-reactive peptide (CRP), white blood cell count, cytokines
Intracellular signalling pathway activation | measured at baseline and after 3 hours of clamp
  Intracellular signalling pathway activation in muscle and fat
Energy expenditure | measured at baseline and after 3 hours of clamp for 15 minutes
  measured by indirect calorimetry
Glucose metabolism | measured at baseline and after 3 hours of clamp
  measured by glucose tracer, calculations of rate of appearance, disappearance and endogenous glucose production
Hormonal changes | measured at baseline and after 3 hours of clamp
  measures of insulin, glucagon, c-peptide and growth hormone
CD163 | 0, 24 and 48 hours after LPS exposure
  measures of CD163 and soluble CD163 (sCD163) after LPS exposure
Fat metabolism | measured at baseline and after 3 hours of clamp
  measured by palmitate tracer, calculating whole body palmitate flux. Measures of free fatty acids.
Urea balance | measured at baseline and after 3 hours of clamp
  measured by urea tracer and urine nitrogen excretion.
Glucose uptake by the forearm | measured at baseline and after 3 hours of clamp
  Arterio-venous balance x blodflow

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Institute for Clinical Medicine
Locations (1):
- Institute for Clinical MEdicine, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No